CLINICAL TRIAL: NCT06975267
Title: The Effectiveness of the Norwegian Version of Second Step Early Learning vs. Free Play on Socio-Emotional Learning in Kindergarten: A Cluster Randomized Controlled Trial Protocol
Brief Title: Social and Emotional Learning in Norwegian Kindergarten
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold University College (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OstfoldUC300802; 353778 (Other Grant/Funding Number: Norwegian Research Council)
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Universal Behavioral Supports
Keywords: Teacher training; second step

STUDY DESIGN:
Intervention Model Description: Cluster randomized controll trial.
Who Masked: Outcomes Assessor
Masking Description: Researchers are masked to the link between participant numbers and assigned arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norwegian version of second step early learning (Experimental): The Norwegian version of the Second Step Early Learning program, in Norwegian called Steg for steg, Småsteg. This is a 28 weeks program divided into five themes which aims to enhance and strengthen children's abilities to learn, show empathy, handle their emotions, friendships, and problem solving.
  Interventions: Behavioral: Norwegian version of Second Step Early Learning
- Free play (Active Comparator): As an active comparator, these children will get the additional time for free play in their kindergartens. The additional time is a reflection of the duration of the program in the intervention group.
  Interventions: Behavioral: Free play

INTERVENTIONS:
Behavioral: Norwegian version of Second Step Early Learning — The interventions is a 28 weeks program divided into five themes. The themes are 1. Skills that promotes learning, 2. Empathy, 3. Managing emotions, 4. Friendship skills and problem solving, and 5. Transitioning to school.
  The intervention consists of daily activities. The guidebook is a central part of the program and provides the kindergarten teachers with practical tools and activities to implement the program in everyday settings. The guidebook includes:
  28 weekly themes: Each week introduces a new theme with related activities and discussion topics.
  Brain-building games: Activities designed to strengthen children's cognitive skills and self-regulation.
  Songs and music: Songs that reinforce the learning of social skills. Parent connections: Information sheets and activities to involve parents in their children's social-emotional development.
  Puppet theatre: The use of hand puppets Dog and Snail to illustrate and discuss feelings and social situations.
  Other Names: Steg for Steg, Småsteg (Norwegian name)
  Arms: Norwegian version of second step early learning
Behavioral: Free play — Control kindergartens will have additional designated playtime consisting of free play for 28 weeks. The checklist for play conditions is defined as when: Time is set aside in the daily kindergarten routine where (1) it is clearly announced or signaled to the children that it is now "free play", (2) it is an absence of requirements for sedentary sitting (unless it is part of the children's play), (3) it is not a situation where children are required to follow instructions (unless it is part of the children's play or general rules in the kindergarten (?)), (4) it is an absence of a pronounced learning outcome or goal with the activities available for the children (beyond what is defined by the children themselves), (5) the children can start and finish activities themselves, and choose what they want to participate in, and (6) adults can join in the game/initiate, but on the children's terms, and the children can choose to leave this game whenever they want.
  Arms: Free play

SUMMARY:
This project evaluates the effectiveness of the Norwegian version of Second Step Early Learning (Småsteg), a program of 28 weeks that emphasizes learning, friendship skills, and managing several strong feelings (e.g., scared, worried, surprised, frustrated, excited), not only anger, on socio-emotional learning (SEL) in kindergartens versus play is a cluster randomized controlled trial. The hypothesis states that Småsteg is superior to play only in improving children's SEL. In the study, 990 children within 66 kindergartens will be recruited and allocated following the randomization at the school level. The primary outcome is based on the Strength and Difficulties Questionnaire (SDQ), which will be answered by parents and teachers at baseline, immediately after the 28 weeks of intervention and then six months after the change to the new school (K1). The secondary outcome is empathy, assessed by the Empathy Questionnaire for Children (EmQue), a parent report-based questionnaire comprising 15 items assessing three domains: emotion contagion, attention to other's feelings, and prosocial actions.

Småsteg could impact the joint attention score, which, in turn, affects the SDQ score. A mobile application (app) will be developed to track children's behaviors via teachers, parents, and children's activities. This study contributes to the scientific understanding of how such interventions can impact SEL and future academic achievement in kindergarten-aged children but also brings insights into mechanisms throughout intervention like Småsteg in early childhood might help the development of SEL, shaping early education policies and practices.

ELIGIBILITY:
Inclusion Criteria:

* All children in the appropriate age group are eligble for inclusion in the study.
* Kindergarten with approximately 15 children or more in the age group are eligble for enrollment.

Exclusion Criteria:

* Kindergartens cannot have implemented the Norwegian version of Second Step Early Learning as an active intervention in their kindergarten for at least the past four years from the start of this study.
* Less than 15 participants in the kindergarten.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Strength and Difficulties Questionnaire (SDQ) | At baseline, after end of intervention (week 29), and after a one year follow-up.
  The primary outcome is based on the Strength and Difficulties Questionnaire (SDQ; Goodman et al., 2003), which will be answered by parents and teachers. SDQ has 25 items and covers five dimensions: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior.

SECONDARY OUTCOMES:
Empathy Questionnaire for Children (EmQue) | At baseline, after end of intervention (week 29), and after a one year follow-up.
  The secondary outcome is empathy, measured by parents using the Empathy Questionnaire for Children (EmQue), which comprises 15 items assessing emotion contagion, attention to others' feelings, and prosocial actions (Reiffe et al., 2010).

OTHER OUTCOMES:
Standardized 1st grade tests in Norwegian and mathematics | At the time of one year follow-up.
  A distal exploratory measure of academic achievement score (last month of the first grade) in reading and math represented by the standardized assessment tests (in Norwegian called Kartleggingsprøver) developed by The Norwegian Directorate for Education and Training (2024).

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Cogo-Moreira, Professor, Principal Investigator — Østfold University College
Locations (1):
- Østfold University College, Halden, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dechsling A, Cipriano C, Bortveit L, Fjermestad KW, Karlsen ABA, Akerbaek TM, Tangen CB, Cogo-Moreira H. Examining the effectiveness of Second Step Early Learning versus free play on socio-emotional learning in kindergarten: a cluster randomized controlled trial protocol. Trials. 2025 Aug 26;26(1):308. doi: 10.1186/s13063-025-09047-7. PMID 40859266